CLINICAL TRIAL: NCT00666120
Title: Assessment of Feeding Tolerance in Infants Fed Cow Milk Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mead Johnson Nutrition (Industry)
Responsible Party: Carol Lynn Berseth, M.D., Mead Johnson
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 3370-6
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Last update posted 2008-04-24 (Estimated); Status verified 2008-04

CONDITIONS: Healthy Term Infants Solely Formula Fed
MeSH Terms: interventions — Iron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Cow's milk based infant formula
  Interventions: Other: Enfamil LIPIL with iron
- 2 (Active Comparator): Partially hydrolyzed cow's milk based infant formula
  Interventions: Other: Good Start Supreme with DHA and ARA

INTERVENTIONS:
Other: Enfamil LIPIL with iron — cow's milk based infant formula
  Arms: 1
Other: Good Start Supreme with DHA and ARA — partially hydrolzed cow's milk protein
  Arms: 2

SUMMARY:
To compare the number of infants who discontinue from study formula due to formula intolerance as documented by the investigator.

Hypothesize there will be no difference between formula groups.

ELIGIBILITY:
Inclusion Criteria:

* Singleton birth
* Term infant at birth
* Birth weight of 2500 g (5 lbs 8 oz) or more
* 4 - 18 days of age at Study Visit 1

Exclusion Criteria:

* History of underlying metabolic or chronic disease or congenital malformation
* Infant switched formulas more than one time between birth and Study Visit 1
* Known feeding problems at Study Visit 1

Ages: 4 Days to 18 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 333 (Actual)
Dates: Start 2005-06; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Number of infants who discontinue from study formula due to formula intolerance as documented by the investigator | 60 days

SECONDARY OUTCOMES:
Infant temperament | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Carol Berseth, MD, Study Director — Mead Johnson Nutrition
Locations (18):
- United States (18):
  - Harvey Pediatrics, Jonesboro, Arkansas
  - Mercy Rogers Pediatric Clinic, Rogers, Arkansas
  - Lovelace Scientific Resources, Santa Ana, California
  - Tampa Bay Medical Research, Clearwater, Florida
  - Children's Medical Association, Tamarac, Florida
  - Children's Health Care, DeKalb, Illinois
  - Welborn Clinic, Evansville, Indiana
  - Fomon Infant Nutrition Unit, Iowa City, Iowa
  - Heartland Research Associates, Wichita, Kansas
  - Pediatrics Clinical Trials Unit, Louisville, Kentucky
  - Pedia Research, Owensboro, Kentucky
  - Arklatex Children's Center, Bossier City, Louisiana
  - Craig Spiegel, MD, Bridgeton, Missouri
  - The Center for Human Nutrition, Omaha, Nebraska
  - Boystown, Omaha, Nebraska
  - Winthrop Pediatric Associates, Mineola, New York
  - Cary Pediatric Center, Cary, North Carolina
  - Collom and Carney Clinic, Texarkana, Texas

REFERENCES:
- [Derived] Berseth CL, Mitmesser SH, Ziegler EE, Marunycz JD, Vanderhoof J. Tolerance of a standard intact protein formula versus a partially hydrolyzed formula in healthy, term infants. Nutr J. 2009 Jun 19;8:27. doi: 10.1186/1475-2891-8-27. PMID 19545360